CLINICAL TRIAL: NCT03521687
Title: An Open-label Pilot Study to Investigate the Efficacy of Apremilast in the Treatment of Central Centrifugal Cicatricial Alopecia (CCCA)
Brief Title: Apremilast in the Treatment of Central Centrifugal Cicatricial Alopecia (CCCA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Saakshi Khattri, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-2386
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Central Centrifugal Cicatricial Alopecia
Keywords: Central centrifugal cicatricial alopecia; open-label pilot study
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Intervention Model Description: This is an open-label study that will enroll 20 subjects with central centrifugal cicatricial alopecia. All subjects will receive apremilast.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Apremilast (Experimental): Patients with CCCA
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — 30 mg BID

SUMMARY:
This is a single-center, open-label clinical study to study the efficacy of apremilast in the treatment of mild to moderate central centrifugal cicatricial alopecia. The investigators hypothesize that the anti-inflammatory properties of apremilast may play a role in the decreasing scalp inflammation in patients with CCCA and may prevent further hair loss and potentially induce hair regrowth in patients with mild to moderate disease.

DETAILED DESCRIPTION:
Central centrifugal cicatricial alopecia (CCCA) is a type of scarring alopecia commonly seen in women of African American descent. The etiology is not completely understood, but CCCA likely results from a combination of hair-grooming practices, a pro-inflammatory state within the hair follicles, and genetic factors. The management of CCCA remains a challenge as there are no published treatment guidelines. Current therapies aim to decrease inflammation in order to prevent further hair loss.

Apremilast, an oral phosphodiesterase-4 inhibitor, has been shown to be effective in the treatment of moderate to severe plaque psoriasis and psoriatic arthropathy. In vitro studies have demonstrated anti-inflammatory properties via inhibition of inflammatory mediators. Therefore, apremilast offers a possible therapeutic option for CCCA. This will be a single-center, open-label clinical study to determine the efficacy of apremilast in the treatment of mild to moderate central centrifugal cicatricial alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, signed and dated informed consent prior to initiating any study-related activities
* Females of African ancestry >18 years of age at the time of screening
* Clinical diagnosis of mild to moderate vertex-predominant CCCA as defined by CHLG stages 1B, 2B, 3B
* Punch biopsy at screening, or punch biopsy of the scalp within six months prior to screening visit, consistent with CCCA
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options.
* Must be in general good health as judged by the Investigator, based on medical history and physical examination. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).

Exclusion Criteria:

* Systemic or intralesional treatment of CCCA for 4 weeks prior to baseline visit, including but not limited to corticosteroids (systemic, intralesional), oral tetracycline antibiotics, and oral anti-inflammatory medications
* Topical corticosteroid or calcineurin inhibitor treatment of CCCA for 2 weeks prior to baseline visit.
* Topical minoxidil for 4 weeks prior to baseline visit.
* Severe or end-stage CCCA with CHLG as defined as CHLG >3
* CCCA with frontal accentuation pattern as defined as CHLG 1A to 5A.
* Diagnosis of other dermatologic diagnosis or condition that, in the opinion of the investigator, would interfere with diagnosis, examination, or treatment of the studied condition (i.e. lichen planopilaris, systemic lupus, cutaneous lupus) or would require treatment with systemic steroids, topical or intralesional steroids on the scalp, or systemic tetracycline antibiotic therapy during the duration of the study.
* Other than the disease under study, any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
* Malignancy or history of malignancy, except for: treated [ie, cured] basal cell or squamous cell in situ skin carcinomas; treated [ie, cured] cervical intraepithelial neoplasia (CIN) or carcinoma in situ of cervix with no evidence of recurrence within the previous 5 years.
* Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.
* Use of systemic immunosuppressive drugs (including, but not limited to, cyclosporine, corticosteroids, mycophenolate mofetil, azathioprine, methotrexate, or tacrolimus) within four weeks prior to Baseline/Randomization (Visit 2).
* Prior history of suicide attempt at any time in the subject's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
* Pregnant or breast feeding.
* Subjects not willing to implement the following suggested hair care practices and/or maintain the same or similar hair style for the duration of study: Shampoo hair every 7 days with a conditioning shampoo; Condition hair every 7 days with a deep or reconstructive conditioner; Towel-dry hair before exposing it to a dryer to minimize excessive heat; Comb hair daily with a wide-toothed comb; gently pass the comb through hair starting from the ends and working your way up to the roots; Avoid heavy pomades and hair oils to scalp; opt for silicone based products or light pomades to hair shafts; Limit use of styling gels; Limit traction-associated hair styles (e.g. tight braids, tight weaves, tight cornrows) as determined by investigator; Avoid chemical or thermal injury to scalp during hair styling process; Chemical relaxer treatments can be used as long as there is no associated scalp injury (i.e. tingling, burning, pain); Maintain the same hair style throughout the study i.e. weave or braids present at baseline must be maintained through the end of the study; weaves or braids may be redone during the study if needed, but should resemble the subject's hair style at baseline, if possible.
* Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamics half-lives, if known (whichever is longer).
* Prior treatment with apremilast
* History of allergy to any component of the IP
* Active substance abuse or a history of substance abuse within 6 months prior to Screening.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female subjects will be enrolled.
Enrollment: 20 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saakshi Khattri, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West Dermatology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with Celgene, who is providing a grant for this study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period from November 2018 to July 2020
Period: Overall Study
Arm/Group | Apremilast
Started | 20
Completed | 15
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Apremilast
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Physician Global Assessment of Improvement (PGA-I)
Description: Mean change in PGA-I at Week 24 compared to Baseline. Trained study personnel will take standardized photographs of the scalp. These photographs will be provided to a panel of three dermatologists with expertise in CCCA, each of whom will review the photographs at these time points. Investigators will assess the improvement in hair loss severity using PGA-I. PGA-I will range from -3 (significant worsening) to 3 (significant improvement).
Time Frame: Week 0 and Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 15
score on a scale | 0.07 (0.51)

2. Secondary Outcome: Mean Change in CCCA Investigator Global Severity Score (IGSS)
Description: Mean change in IGSS at Week 24 compared to Baseline. Treatment response will be considered no change or improvement in IGSS. CCCA Investigator Global Severity Score (IGSS) assess subjects on a scale of 0 (no hair loss) to 6 (severe CCCA, e.g. >75% involvement of vertex).
Time Frame: Week 0 and Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 15
score on a scale | -0.31 (0.65)

3. Secondary Outcome: Mean Change in Central Hair Loss Grade (CHLG)
Description: Mean change in CHLG at Week 24 compared to Baseline. Degree of severity of hair loss is graded on a 6-point visual scale (pattern 0: no hair loss, pattern 1-2: mild hair loss, pattern 3-5: more severe hair loss).
Time Frame: Week 0 and week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 15
score on a scale | -0.44 (0.86)

4. Secondary Outcome: Mean Change in Subject Visual Analog Scale (VAS) of Hair Loss Severity
Description: Mean change in VAS at Week 24 compared to Baseline. The VAS is a numerical scale used to assess patients' perception of hair loss severity. The evaluation is a 10cm long line on which the subjects indicate the severity of their condition from "0" (complete loss of hair in affected area - ie no visible hairs on central scalp) to "10" (full growth/regrowth in affected area-ie no visible hair loss on central scalp).
Time Frame: Week 0 and Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 15
score on a scale | -1.94 (1.86)

5. Secondary Outcome: Mean Change in Subject Global Assessment of Improvement
Description: Mean change in PaGA-I at Week 24 as compared to Baseline. PaGA-I will range from -3 (significant worsening) to 3 (significant improvement).
Time Frame: Week 0 and Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 15
score on a scale | 1 (1.45)

6. Secondary Outcome: Change in Subject Rating of Symptom Severity Questionnaire (NRS)
Description: Change in NRS at Week 24 as compared to Baseline. Subjects will complete a symptom severity questionnaire consisting of 3 numeric rating scales (NRS) measuring severity of pruritus, burning, and pain. The NRS will range from 0 (no symptoms) to 10 (severe symptoms). Patients indicate the intensity of each symptom (pruritus, burning, or pain) by choosing a number from 0 to 10 that corresponds to the severity of that symptom.
Time Frame: Week 0 and Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 15
score on a scale | 0.94 (3.99)

7. Secondary Outcome: Mean Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score
Description: Mean change in DLQI total score at Week 24 as compared to Baseline. DLQi is a 10-item questionnaire, each question is scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
Time Frame: Week 0 and Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 15
score on a scale | -2.18 (3.79)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Apremilast
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 19/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apremilast (N=20)
Nausea (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 3
Reflux (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 5
Loose stools (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 3
Depression (Psychiatric disorders) | 3
Decreased appetite (General disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Weight Loss (General disorders) | 3
Common cold (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 3
Tiredness (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Increased bowel movements (Gastrointestinal disorders) | 5
Covid like illness (Infections and infestations) | 3
Increased hair loss (Skin and subcutaneous tissue disorders) | 2
Nasal congestion (General disorders) | 1
Cracked tooth (General disorders) | 1
Anxiety (Psychiatric disorders) | 1
Lower back muscle strain (Musculoskeletal and connective tissue disorders) | 1
left knee pain (Musculoskeletal and connective tissue disorders) | 1
Itchy scalp (Skin and subcutaneous tissue disorders) | 1
Seasonal allergies (General disorders) | 1
Sinus headache (General disorders) | 1
Hair breakage (Psychiatric disorders) | 1
Sinusitis (General disorders) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Worsening urticaria (Skin and subcutaneous tissue disorders) | 1
Intention tremor (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Subjective PIH (Skin and subcutaneous tissue disorders) | 1
Hyperactivity (Psychiatric disorders) | 1
Abnormal mammogram (Reproductive system and breast disorders) | 1
Post nasal drip (General disorders) | 1
Irregular periods (Reproductive system and breast disorders) | 1
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 1
Eye Infection (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT03521687/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT03521687/SAP_001.pdf